CLINICAL TRIAL: NCT03399643
Title: Non-Interventional Study To Investigate The Effectiveness Of Atezolizumab Under Real-World Conditions In Patients With Inoperable Locally-Advanced Or Metastatic Urothelial Carcinoma Of The Urinary Tract (Announce)
Brief Title: A Study to Investigate The Effectiveness Of Atezolizumab In Patients With Inoperable Locally-Advanced Or Metastatic Urothelial Carcinoma Of The Urinary Tract (Announce)
Acronym: Announce
Status: Terminated | Type: Observational
Why Stopped: Tecentriq label restriction for first line limited the patient population and scientific question could not be answered in an appropriate time.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39704
Record Dates: First submitted 2017-12-19; First posted 2018-01-16 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is administered via IV 1200 mg every 3 weeks

SUMMARY:
The objective of this study is to investigate the effectiveness of Atezolizumab with a primary focus on the overall survival (OS) rate at 2 years and secondary focuses on quality of life (QoL) and the sequence of treatment in mUC patients. Furthermore, this study aims at collecting data on safety of Atezolizumab and on the reason for cisplatin-ineligibility

ELIGIBILITY:
Inclusion Criteria:

* Metastatic UC (Urothelial Carcinoma) including cancers of the renal pelvis, ureters, urinary bladder, and urethra
* Will be receiving atezolizumab for the treatment of inoperable locally-advanced or metastatic UC, per the decision of the treating physician
* Have adequate hematologic and end-organ functions
* Have had no prior palliative chemotherapy for inoperable locally-advanced or metastatic UC and are clinically ineligible ("unfit") for cisplatin-based chemotherapy

Exclusion Criteria:

* Have received prior immune checkpoint therapy
* Are pregnant or breastfeeding
* Are included in any other trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients ineligible for palliative cisplatin-based chemotherapy or who received prior adjuvant/ neoadjuvant chemotherapy or chemo radiation with a treatment-free interval more than 12 months (1L)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Overall Survival Rate (OS rate) | 2 years

SECONDARY OUTCOMES:
Median Overall Survival (OS) | Initiation of study treatment until death or end of study, approximately 4 years
Median Progression Free Survival (PFS) | Initiation of study treatment to first measured disease progression, through end of study (approximately 4 years)
Percentage of participants with adverse events | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- Germany (32):
  - Praxis Dr.med. Wolfgang Hölzer, Berlin
  - Urologie Schlosscarree, Braunschweig
  - Urologische Praxis Dr. Krieger, Chemnitz
  - Zeisigwaldkliniken Bethanien, Chemnitz
  - St. Georg Klinikum Eisenach GmbH, Eisenach
  - St. Franziskus-Hospital; Malteser Krankenhaus; Medizinische Klinik I, Flensburg
  - Klinikum Frankfurt Höchst GmbH; Klinik Innere Medizin 3 - Hämatologie, Onkologie, Palliativmedizin, Frankfurt am Main
  - Dres.Jochen Wilke und Harald Wagner, Fürth
  - Krankenhaus Martha-Maria Halle-Dölau, Klinik für Urologie, Halle
  - Urologische Praxis Michael Steinacker, Halle
  - Asklepios Klinik Altona, Abteilung für Urologie, Hamburg
  - Onkologische Praxis in Heidenheim, Heidenheim
  - St. Bernward-Krankenhaus, Hildesheim
  - Onkologische Praxis Landshut, Landshut
  - Gemeinschaftspraxis; Onkologisches Zentrum Lebach; Caritas Krankenhaus Lebach, Lebach
  - ÜBAG MVZ Mitte / MVZ Delitzsch GmbH, Standort Leipzig, Leipzig
  - Sankt Elisabeth Krankenhaus; Urlogische Abt., Leipzig
  - Drk Krankenhaus Luckenwalde, Luckenwalde
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Urologie, Lübeck
  - Urologikum Lübeck, Lübeck
  - Urologischen Praxis in Lüneburg, Lüneburg
  - Medizinische Fakultät Mannheim, Universitätsklinikum Mannheim, Klinik für Urologie, Mannheim
  - Praxis Markkleeberg, Markkleeberg
  - Mühlenkreiskliniken; Johannes Wesling Klinikum Minden; Klinik für Hämatologie, Onkologie und Pallia., Minden
  - Städt.Kliniken München GmbH Klinikum Bogenhausen, München
  - Praxis Dr. Uhlig, Naunhof, Naunhof
  - Brüderkrankenhaus St. Josef Paderborn, Klinik für Hämatologie/Onkologie, Paderborn
  - Praxis für Hämatologie & Onkologie, Saarbrücken
  - MVZ für Hämatologie, Onkologie, Strahlentherapie und Palliativmedizin -; Klinik Dr. Hancken, Stade
  - Krankenhaus der Barmherzigen Brüder Trier; Innere Medizin I, Hämatologie / Internistische Onkologie, Trier
  - Urologische Praxis, Wedel
  - Gemeinschaftspraxis für Hämatologie und Onkologie Westerstede Aurich Rhauder, Westerstede